CLINICAL TRIAL: NCT00236821
Title: Multicenter, Double-Blind Randomized Study to Compare the Safety and Efficacy of Levofloxacin 750 mg Once Daily for Five Days vs. Levofloxacin 500 mg Once Daily for 10 Days in the Treatment of Mild to Severe Community-Acquired Pneumonia in Adults
Brief Title: A Study to Compare the Safety and Effectiveness of 2 Doses of Levofloxacin Given for Different Time Periods in Patients With Pneumonia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: PriCara, Unit of Ortho-McNeil, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR005554
Record Dates: First submitted 2005-10-07; First posted 2005-10-12 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2010-04

CONDITIONS: Pneumonia
Keywords: respiratory tract diseases; pneumonia; levofloxacin; community-acquired pneumonia; lung diseases; quinolones
MeSH Terms: conditions — Pneumonia; Respiratory Tract Diseases; Community-Acquired Pneumonia; Lung Diseases | interventions — Levofloxacin

INTERVENTIONS:
Drug: levofloxacin

SUMMARY:
The purpose of this study is to evaluate the effectiveness and safety of two antibiotic regimens in the treatment of community-acquired pneumonia in non-hospitalized adult patients. A 5-day course of 750 milligrams of levofloxacin given once daily will be compared to a 10-day course 500 milligrams of levofloxacin given once daily.

DETAILED DESCRIPTION:
Levofloxacin is an antibiotic that is approved by the FDA for the treatment of sinusitis, chronic bronchitis, skin infections, urinary tract infections, and community-acquired pneumonia. This multicenter, double-blind (neither the patient nor the study doctor will know the dose of levofloxacin being administered) study evaluates the effectiveness and safety of two antibiotic regimens in the treatment of community-acquired pneumonia in adult patients. A 5-day course of 750 milligrams of levofloxacin given once daily will be compared to a 10-day course 500 milligrams of levofloxacin given once daily. Patients receive levofloxacin by mouth or through a vein depending on the severity of their pneumonia. Patients are assessed after 3 days of treatment; treatment is discontinued if no significant improvement is noted. Patients showing signs of improvement continue in the study, with assessments on study days 12-16, and 17-21 (posttherapy visits), and 31-38 (poststudy visit). Effectiveness is assessed by measuring the ability of the study drug to eliminate bacteria causing pneumonia and to reduce the signs and symptoms of pneumonia. Chest x-rays and laboratory tests for presence of bacteria are performed during the study. Safety evaluations (incidence of adverse events, physical examinations, laboratory tests) are performed throughout the study. The study hypothesis is that levofloxacin administered at a higher dose for a shorter duration is at least as effective as levofloxacin administered at a lower dose for a longer duration in the treatment of community-acquired pneumonia and is generally well-tolerated.

Levofloxacin, 500 milligrams (mg) by mouth or through vein daily for 10 days or 750 mg by mouth or slowly through a vein daily for 5 days

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of community-acquired pneumonia as follows: clinical signs and symptoms of a lower respiratory tract infection and chest-x-ray findings consistent with pneumonia within 24 hours before entry into the study
* At least one of the following: abnormal temperature (high or low) or abnormal white blood cell count
* Previous antibiotic treatment <= 24 hours or, if the duration of treatment was >= 72 hours and that therapy failed based on at least 2 of the following: fever within 12 hours of entry into the study, chest x-ray findings have worsened compared to the initial chest-x-ray, white blood cell count is significantly increased, respiratory rate higher than at the start of treatment and >= 20 breaths per minute or need for supplemental oxygen if not previously needed
* Patients whose infection is acquired in the community or, if in a nursing home, who had been living there < 14 days
* Fine Class (rating scale used to assess patients' overall condition which includes information such as age, gender, other diseases, physical examination and laboratory findings) score <= 130 upon admission (patients with Fine Class scores > 70 but < = 130 must initially be hospitalized
* Patients with scores of <= 70 may be treated as outpatients or hospitalized at the discretion of the investigator)

Exclusion Criteria:

* Pneumonia known or suspected to be due to a bacteria resistant to levofloxacin
* Previous allergic or serious reaction to or failed therapy with levofloxacin or similar drugs
* Life expectancy < 72 hours
* Hospitalized within 2 weeks before entry in the study or within 1 month before entry in the study if treated with antibiotics
* Pneumonia acquired in a hospital
* Cystic fibrosis or other lung disorders
* Receiving chronic steroid treatment
* Received assistance from a machine to breathe within the previous month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 530 (Actual)
Dates: Start 2001-03; Study Completion 2002-06 (Actual)

PRIMARY OUTCOMES:
Clinical response rates based on signs and symptoms at posttherapy visit.

SECONDARY OUTCOMES:
Microbiologic eradication rates at posttherapy visit; Clinical response rates (chest x-ray findings and signs/symptoms) and microbiologic eradication rates at poststudy; Incidence of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research and Development, L.L.C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Result] Dunbar LM, Wunderink RG, Habib MP, Smith LG, Tennenberg AM, Khashab MM, Wiesinger BA, Xiang JX, Zadeikis N, Kahn JB. High-dose, short-course levofloxacin for community-acquired pneumonia: a new treatment paradigm. Clin Infect Dis. 2003 Sep 15;37(6):752-60. doi: 10.1086/377539. Epub 2003 Aug 28. PMID 12955634
- See also: A study to compare the safety and effectiveness of 2 doses of levofloxacin given for different time periods in patients with pneumonia — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=663&filename=CR005554_CSR.pdf